CLINICAL TRIAL: NCT01517932
Title: Effects of Dexmedetomidine on Stress Response and Postoperative Analgesia in Patients Undergoing Thoracotomy During Anesthesia Recovery Period
Brief Title: Effects of Dexmedetomidine on Stress Response and Postoperative Analgesia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fang Luo (Other)
Responsible Party: Sponsor-Investigator, Fang Luo, Department of Anesthesiology, Tongji Hospital, Tongji medical college, Huazhong University of science and Technology, Huazhong University of Science and Technology
Organization: Huazhong University of Science and Technology (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: TJMU-A-201106
Record Dates: First submitted 2012-01-22; First posted 2012-01-25 (Estimated); Last update posted 2013-03-20 (Estimated); Status verified 2013-03

CONDITIONS: Restlessness; Pain
MeSH Terms: conditions — Psychomotor Agitation; Pain | interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group-DEX (Experimental): Patients in this arm received dexmedetomidine 0.2 microgram per kg i.v. during 10 minutes 1 hour before the end of surgery
  Interventions: Drug: dexmedetomidine
- Group-PLB (Placebo Comparator): Patients in this arm received saline placebo 0.05 ml per kilogram i.v. during 10 minutes 1 hour before the end of surgery
  Interventions: Drug: saline placebo

INTERVENTIONS:
Drug: dexmedetomidine — In this arm,midazolam(0.03-0.05mg/kg), propofol(1.5-2.5mg/kg),sufentanil(0.6-0.82μg/kg )and rocuronium(0.8-1.0mg/kg) were used in anesthesia induction.
  Anaesthesia was maintained with propofol（4-6mg kg-1h-1），remifentanil (0.1-0.2 μg kg-1 min-1）and sevoflurane（1%).Propofol was titrated to maintain intraoperative Narcotrend values between 20 and 46.
  Patients in this arm received dexmedetomidine 0.2μg/kg i.v. during 10 minutes 1 hour before the end of surgery
  Arms: Group-DEX
Drug: saline placebo — In this arm,midazolam(0.03-0.05mg/kg), propofol(1.5-2.5mg/kg),sufentanil(0.6-0.82μg/kg )and rocuronium(0.8-1.0mg/kg) were used in anesthesia induction.
  Anaesthesia was maintained with propofol（4-6mg kg-1h-1），remifentanil (0.1-0.2 μg kg-1 min-1）and sevoflurane（1%).Propofol was titrated to maintain intraoperative Narcotrend values between 20 and 46.
  Patients in this arm received saline placebo of the same volume i.v. during 10 minutes 1 hour before the end of surgery
  Arms: Group-PLB

SUMMARY:
Dexmedetomidine is a highly selective α2 adrenoreceptor agonist approved by the US FDA for short-term postoperative sedation and analgesia.It can also reduce the stress response without respiratory depression.

In this prospective, randomized, double-blind, placebo-controlled study，we gave dexmedetomidine or saline placebo 1h before operations were over and assessed the effects of dexmedetomidine on stress response and postoperative analgesia in patients undergoing thoracotomy during anesthesia recovery period.

DETAILED DESCRIPTION:
Dexmedetomidine can significantly reduce the emergence agitation and postoperative pain in patients who received chest surgery

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anaesthesiologists Physical Status (ASA-PS) I or II
* undergoing selective thoracotomy
* weight between 45 and 75kg
* operation time 2-4 hours

Exclusion Criteria:

* history of neurologic disease
* history of chronic analgesics intake
* history of allergic reactions to the experimental durgs
* history of renal insufficiency
* history of hepatic dysfunction
* history of coagulation disorders
* women in lactation
* participating in other studies

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-06; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Emergence agitation | during 0-3 postoperative hours
  Emergence agitation was assessed by the highest restlessness score（RS）during 0-3 postoperative hours

SECONDARY OUTCOMES:
Postoperative pain at rest | At 1,3 postoperative hours
  The patients were instructed to give the number that represented the pain level at rest by using visual analogue scale（VAS）and prince-henry score
dosage Dosage of analgesics | during 3 postoperative hours
Recovery time | At the moment of the eyes opend when calling the names
Postoperative sedation | at 0,1,3 postoperative hours
  It was assessed by Ramsay Sedation Score(RSS)
Extubation time | at the moment of extubation
Breathing recovery time | when autonomous respiration recovered

CONTACTS AND LOCATIONS:
Overall Officials: Fang Luo, MD.PhD, Study Director — Department of Anaesthesiology, Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, 1095 Jiefang Avenue, Wuhan 430030, China